CLINICAL TRIAL: NCT02307630
Title: PET Imaging of Solid Tumors Using 124I-Humanized 3F8: A Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-147
Record Dates: First submitted 2014-11-20; First posted 2014-12-04 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Melanoma; Neuroblastoma; Sarcoma
Keywords: 124I-Humanized 3F8; PET Imaging; 13-147
MeSH Terms: conditions — Melanoma; Neuroblastoma; Sarcoma

ARMS (1):
- PET Imaging using 124I-Humanized 3F8 (Experimental): 124I-hu3F8 at a dose of 3mCi/m2 (with a maximum dose of 5mCi) will be injected IV. 124I-hu3F8 PET/CT scans will be performed at approximately 2-4 hours, 18-26hours, 48-72 hours and 96-144 hours after injection of 124I-hu3F8. A low dose CT scan will be obtained with each PET scans. PET/CT scan images will be analyzed to determine biodistribution of 124I-hu3F8 and to determine dosimetry to organs and sites of disease. Comparison of tumor targeting and tumor dosimetry will be made between the two cohorts of patients: (a) NB and (b) other solid tumors. Blood will be drawn where feasible at multiple time points: approximately 0h, 0.5h, 1h, 2h, 4-8h, 24h, 48h, 96h and 120h-144h after injection of 124I-hu3F8 and radioactivity measured to determine pharmacokinetics of 124I-hu3F8.
  Interventions: Biological: 124I-Humanized 3F8

INTERVENTIONS:
Biological: 124I-Humanized 3F8

SUMMARY:
The purpose of this study is to find out how an antibody called Hu3F8 travels through the body and to tumors. Antibodies, like Hu3F8, are proteins that help attack tumors or fight infections. Antibodies can be made by your own body or in a laboratory. The target of an antibody is called an antigen; antibodies fit their antigen like a lock fits a key.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of neuroblastoma must meet both of the following criteria:

  * Diagnosis confirmed by histological assessment by MSKCC Department of pathology or by the presence of BM metastases PLUS elevated urinary catecholamines
  * Relapsed or refractory stage 4 disease or relapsed or refractory stage MYCN-amplified 2B or 3 disease.
  * Patients with tumors other than neuroblastoma must meet both the following criteria:
  * Have one of the following diagnoses (these tumors are known to express GD2 on cell surface):
  * Melanoma
  * Osteogenic sarcoma
  * Leiomyosarcoma
  * Ewing sarcoma
  * Liposarcoma
  * Fibrosarcoma
  * Malignant fibrous histiocytoma
  * Spindle cell sarcoma
  * Small cell lung cancer
  * Medulloblastoma metastatic to extracranial sites
  * Paraganglioma
  * Have refractory or relapsed or metastatic disease
  * Patients with solid tumors with diagnoses OTHER than neuroblastoma or those listed above will be eligible if they meet both of the following criteria:
  * Immunohistochemical demonstration of GD2 expression on cell surface (Tumor assessment by immunohistochemistry is required for this group of patients)
  * Have refractory or relapsed disease or metastatic disease. All patients must have measurable or evaluable disease
  * Age 3-90 years
  * Prior treatment with anti-GD2 monoclonal antibody is permitted only if human anti-human antibody titer is ≤1300 assay developed by Dr. Nai-Kong Cheung.
  * Negative serum pregnancy test in women of childbearing potential
  * Women of child-bearing potential must be willing to practice an effective method of birth control while on study
  * Signed informed consent indicating awareness of the investigational nature of this study.

Exclusion Criteria:

* Existing major organ dysfunction > grade 2, with the exception of myelosuppression (neutrophil count > or = 500/μl and platelet count > or = 25,000/μl are acceptable) and hearing loss.

  * Acute life threatening infection
  * Requirement for sedation for PET/CT scans
  * Pregnant women or women who are breast-feeding.
  * Inability to comply with protocol requirements.
  * Hypersensitivity to potassium iodide or Lugols products
  * Prior development of positive human antimouse antibody response (HAMA) or human antihuman antibody response (HAHA)
  * Positive human anti-hu3F8 antibody titer.

Ages: 3 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
radioactivity measured to determine pharmacokinetics of 124I-hu3F8 | 2 years
  Following 124I-hu3F8 administration, upon completion of normal saline flush, blood will be drawn for pharmacokinetic studies at the following time points: 0h, 0.5h, 1h, 2h, 4-8h, 24h, 48h, 96h and 120-144 h.after injection of 124I-hu3F8 and radioactivity measured to determine pharmacokinetics of 124I-hu3F8.

SECONDARY OUTCOMES:
PET/CT scan images will be analyzed to determine bio distribution of 124I-hu3F8 | 2 years
  124I-hu3F8 will be injected IV followed by PET/CT scans at serial timepoints PET/CT scan images will be analyzed to determine biodistribution of 124I-hu3F8

CONTACTS AND LOCATIONS:
Overall Officials: Shakeel Modak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/